CLINICAL TRIAL: NCT03653221
Title: Developing of Virtual Reality Based Neurologic Examination Teaching Tool(VRNET)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Other
Other Study IDs: 4-2018-0665
Record Dates: First submitted 2018-08-27; First posted 2018-08-31 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Medical Students

STUDY DESIGN:
Intervention Model Description: 1. standardized patients with VRNET
  2. standardized patients
Who Masked: Investigator, Outcomes Assessor
Masking Description: investigator, outcome assessors will be blinded for group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standardized patients with VRNET (Experimental): The medical students examine the standardized patients who have neurological deficits which presented by VRNET.
  Interventions: Other: Standard patients with VRNET
- standardized patients (Placebo Comparator): The medical students examine the standardized patients who have neurological deficits which presented by words or pictures.
  Interventions: Other: standard patients

INTERVENTIONS:
Other: Standard patients with VRNET — In group of standard patients with VRNET, the medical students examine the standard patient of neurologic deficits. When they examine, they get some information of neurologic signs via the VRNET which presents neurologic deficits directly by alternating facial expressions. The students should interpret that signs to have a diagnosis.
  Arms: standardized patients with VRNET
Other: standard patients — In group of standard patients, those neurological deficits are presented only by words or pictures which are not realistic.
  Arms: standardized patients

SUMMARY:
The purpose of this study is to evaluate the effect of the virtual reality based neurologic examination teaching tool(VRNET) for medical students. VRNET is a new teaching tool for neurologic examinations by offering different neurologic signs of the face, with which medical students can experience more realistic patients.

ELIGIBILITY:
Inclusion Criteria:

* 4th grade medical students of emergency medicine clerkship who agree with participation on this study.

Exclusion Criteria:

* Disagree with participation on this study.
* Who are absent the last day of clerkship.

Ages: 23 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 95 (Actual)
Dates: Start 2019-03-18 (Actual); Primary Completion 2019-07-12 (Actual); Study Completion 2019-07-12 (Actual)

PRIMARY OUTCOMES:
Neurologic physical exam(NPE) score | after 2 weeks clinical clerkship rotation.
  NPE score is consist of 6 neurologic examination parts; cranial nerve, motor, sensory, cerebellar function, gait. Each part has 1 points, so NPE score ranges from 0 to 6. NPE score of students is evaluated by neurologist viewing video clips which recorded during the last day of 2 weeks clerkship rotation.

SECONDARY OUTCOMES:
Satisfaction of students for VRNET | after 2 weeks clinical clerkship rotation.
  Satisfaction of VRNET are evaluated by students' answer to the question below with Likert scale (0 to 5) after completion examination of standard patient.
  "I am satisfied with VRNET for neurologic examination training. 0 (not at all)---1----2----3-----4-----5 (very helpful)"
Reality of VRNET by students | after 2 weeks clinical clerkship rotation.
  Reality of VRNET are evaluated by students' answer to the question below with Likert scale (0 to 5) after completion examination of standard patient.
  "VRNET is very realistic. 0 (not at all)---1----2----3-----4-----5 (very realistic)"
Evaluation of students by standardized patients | after 2 weeks clinical clerkship rotation.
  Evaluation of students by standard patients is also using Likert scale (0 to 5) based on the pre-made check lists.
  "How do you feel as a standard patient that the student did good job?" 0 (not at all)---1----2----3-----4-----5 (very competent)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of emergency medicine, Yonsei University College of Medicine, Seoul, Korea, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No